CLINICAL TRIAL: NCT00162240
Title: A Phase 3, Randomized, Double-blind, Placebo Controlled, Multicenter Trial to Evaluate the Safety and Efficacy of BMS-298585 in Combination With Metformin Therapy in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control on Metformin Therapy Alone
Brief Title: PPAR - Combination With Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV168-022
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Diabetes Mellitus
Keywords: Metabolics Diabetes New Onset
MeSH Terms: conditions — Diabetes Mellitus | interventions — muraglitazar

INTERVENTIONS:
Drug: Muraglitazar

SUMMARY:
A Phase 3, Randomized, Double-blind, Placebo Controlled, Multicenter Trial to Evaluate the Safety and Efficacy of BMS-298585 in Combination with Metformin Therapy in Subjects with Type 2 Diabetes Who Have Inadequate Glycemic Control on Metformin Therapy Alone

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* HbA1c > - 7.0% and < - 10.0 %
* Mean serum triglyceride < - 600 mg/dL
* Body mass index < - 41 kg/m2
* Fasting c-peptide > - 1.0 ng/mL

Exclusion Criteria:

* History of myocardial infarction (MI)
* coronary angioplasty or bypass graft(s)
* valvular disease or repair
* unstable angina pectoris
* transient ischemic attack (TIA), cerebrovascular attack, or cerebrovascular accident (CVA) within 6 months
* Congestive heart failure NYHA Class III and IV
* Uncontrolled hypertension
* History of renal disease, peripheral vascular disease (PVD), pulmonary disease, gastrointestinal disease, active liver disease or endocrine disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534
Dates: Start 2003-06; Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
compare change from baseline in HbA1c after 24 weeks of treatment with muraglitazar + metformin vs placebo + metformin

SECONDARY OUTCOMES:
change in FPG from basline to W24, proportion of subjects receiving therapeutic response at W24, percent change of fasting lipid levels from baseline to W11/12, change in hs-CRP from baseline to W24

CONTACTS AND LOCATIONS:
Locations (203):
- United States (108):
  - Local Institution, Anniston, Alabama
  - Local Institution, Birmingham, Alabama
  - Local Institution, Haleyville, Alabama
  - Local Institution, Mobile, Alabama
  - Local Institution, Mesa, Arizona
  - Local Institution, Phoenix, Arizona
  - Local Institution, Tucson, Arizona
  - Local Institution, Fayette, Arkansas
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Concord, California
  - Local Institution, Fountain Valley, California
  - Local Institution, La Jolla, California
  - Local Institution, Los Angeles, California
  - Local Institution, Los Gatos, California
  - Local Institution, Mission Viejo, California
  - Local Institution, Pasadena, California
  - Local Institution, Rolling Hills Estate, California
  - Local Institution, Roseville, California
  - Local Institution, San Diego, California
  - Local Institution, Spring Valley, California
  - Local Institution, Walnut Creek, California
  - Local Institution, Colorado Springs, Colorado
  - Local Institution, Denver, Colorado
  - Local Institution, Littleton, Colorado
  - Local Institution, Loveland, Colorado
  - Local Institution, Wheat Ridge, Colorado
  - Local Institution, New Britain, Connecticut
  - Local Institution, Newark, Delaware
  - Local Institution, Wilmington, Delaware
  - Local Institution, Chipley, Florida
  - Local Institution, Cooper City, Florida
  - Local Institution, Kissimmee, Florida
  - Local Institution, Melbourne, Florida
  - Local Institution, Miami, Florida
  - Local Institution, New Port Richey, Florida
  - Local Institution, Ocala, Florida
  - Local Institution, Orlando, Florida
  - Local Institution, Winter Park, Florida
  - Local Institution, Columbus, Georgia
  - Local Institution, Dunwoody, Georgia
  - Local Institution, Honolulu, Hawaii
  - Local Institution, Overland Park, Kansas
  - Local Institution, Shawnee Mission, Kansas
  - Local Institution, Wichita, Kansas
  - Local Institution, Louisville, Kentucky
  - Local Institution, Richmond, Kentucky
  - Local Institution, Slidell, Louisiana
  - Local Institution, Chester, Maryland
  - Local Institution, Silver Spring, Maryland
  - Local Institution, Ayer, Massachusetts
  - Local Institution, Springfield, Massachusetts
  - Local Institution, Sudbury, Massachusetts
  - Local Institution, Lansing, Michigan
  - Local Institution, Arden Hills, Minnesota
  - Local Institution, Gulfport, Mississippi
  - Local Institution, Olive Branch, Mississippi
  - Local Institution, Rolling Fork, Mississippi
  - Local Institution, City of Saint Peters, Missouri
  - Local Institution, Excelsior Springs, Missouri
  - Local Institution, Kansas City, Missouri
  - Local Institution, Springfield, Missouri
  - Local Institution, St Louis, Missouri
  - Local Institution, Omaha, Nebraska
  - Local Institution, Toms River, New Jersey
  - Local Institution, Albuquerque, New Mexico
  - Local Institution, Buffalo, New York
  - Local Institution, New Hyde Park, New York
  - Local Institution, West Seneca, New York
  - Local Institution, Westfield, New York
  - Local Institution, Charlotte, North Carolina
  - Local Institution, Durham, North Carolina
  - Local Institution, Greensboro, North Carolina
  - Local Institution, Greenville, North Carolina
  - Local Institution, Hickory, North Carolina
  - Local Institution, High Point, North Carolina
  - Local Institution, Huntersville, North Carolina
  - Local Institution, Salisbury, North Carolina
  - Local Institution, Wilmington, North Carolina
  - Local Institution, Winston-Salem, North Carolina
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Tulsa, Oklahoma
  - Local Institution, Corvallis, Oregon
  - Local Institution, Eugene, Oregon
  - Local Institution, Hillsboro, Oregon
  - Local Institution, Portland, Oregon
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Warminster, Pennsylvania
  - Local Institution, Cranston, Rhode Island
  - Local Institution, Duncan, South Carolina
  - Local Institution, Greer, South Carolina
  - Local Institution, Simpsonville, South Carolina
  - Local Institution, Bristol, Tennessee
  - Local Institution, Kingsport, Tennessee
  - Local Institution, Memphis, Tennessee
  - Local Institution, Dallas, Texas
  - Local Institution, Houston, Texas
  - Local Institution, Irving, Texas
  - Local Institution, Lake Jackson, Texas
  - Local Institution, Lubbock, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Salt Lake City, Utah
  - Local Institution, Springfield, Virginia
  - Local Institution, Virginia Beach, Virginia
  - Local Institution, Olympia, Washington
  - Local Institution, Renton, Washington
  - Local Institution, Spokane, Washington
  - Local Institution, Milwaukee, Wisconsin
- Argentina (5):
  - Local Institution, Bahía Blanca, Buenos Aires
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Buenos Aires, Buenos Aires F.D.
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Mendoza, Mendoza Province
- Australia (6):
  - Local Institution, Canberra, New South Wales
  - Local Institution, Sydney, New South Wales
  - Local Institution, Wollongong, New South Wales
  - Local Institution, Brisbane, Queensland
  - Local Institution, Meadowbrook, Queensland
  - Local Institution, Perth, Western Australia
- Brazil (3):
  - Local Institution, Curitiba, Paraná
  - Local Institution, Belém, Pará
  - Local Institution, Porto Alegre, Rio Grande do Sul
- Canada (19):
  - Local Institution, Calgary, Alberta
  - Local Institution, Coquitlam, British Columbia
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Manuels, Newfoundland and Labrador
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Halifax, Nova Scotia
  - Local Institution, Oakville, Ontario
  - Local Institution, Ottawa, Ontario
  - Local Institution, Thornhill, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Chicoutimi, Quebec
  - Local Institution, Fleurimont, Quebec
  - Local Institution, Granby, Quebec
  - Local Institution, Laval, Quebec
  - Local Institution, Longueuil, Quebec
  - Local Institution, Montreal, Quebec
  - Local Institution, Pointe-Claire, Quebec
  - Local Institution, Sherbrooke, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- France (8):
  - Local Institution, Albens
  - Local Institution, Broglie
  - Local Institution, Chartres
  - Local Institution, Fabrègues
  - Local Institution, Gémenos
  - Local Institution, Husseren-Wesserling
  - Local Institution, Labarthe-sur-Lèze
  - Local Institution, Rosiers-d'Égletons
- Mexico (8):
  - Local Institution, Durango, Durango
  - Local Institution, Tijuana, Estado de Baja California
  - Local Institution, León, Guanajuato
  - Local Institution, Distrito Federal, Mexico City
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Cuernavaca, Morelos
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Mérida, Yucatán
- Peru (2):
  - Local Institution, Arequipa, Arequipa
  - Local Institution, Lima, Lima Province
- Puerto Rico (5):
  - Local Institution, Añasco
  - Local Institution, Carolina
  - Local Institution, Guaynabo
  - Local Institution, Ponce
  - Local Institution, Rio Piedras
- Local Institution, Seoul, South Korea
- Sweden (17):
  - Local Institution, Ängelholm
  - Local Institution, Bjuv
  - Local Institution, Enskede
  - Local Institution, Farsta
  - Local Institution, Gothenburg
  - Local Institution, Helsingborg
  - Local Institution, Jarfalla
  - Local Institution, Landskrona
  - Local Institution, Leksand
  - Local Institution, Linköping
  - Local Institution, Malmo
  - Local Institution, Ödeshög
  - Local Institution, Sävedalen
  - Local Institution, Sjuntorp
  - Local Institution, Stockholm
  - Local Institution, Trollhättan
  - Local Institution, Vällingby
- United Kingdom (21):
  - Local Institution, Carrickfergus, Antrim
  - Local Institution, Soham, Cambridgeshire
  - Local Institution, Doncaster, Derbyshire
  - Local Institution, Paignton, Devon
  - Local Institution, Bangor, Down
  - Local Institution, Downpatrick, Down
  - Local Institution, Bexhill-on-Sea, East Sussex
  - Local Institution, High Valleyfield, Fife
  - Local Institution, Sunbury-on-Thames, Greater London
  - Local Institution, Aldershot, Hampshire
  - Local Institution, Glasgow, Lanarkshire
  - Local Institution, Blackpool, Lancashire
  - Local Institution, Farnworth, Lancashire
  - Local Institution, Harrow, Middlesex
  - Local Institution, Doncaster, North Yorkshire
  - Local Institution, Hastings, Sussex
  - Local Institution, Atherstone, Warwickshire
  - Local Institution, Nuneaton, Warwickshire
  - Local Institution, Bath, Wiltshire
  - Local Institution, Inkberrow, Worcestershire
  - Local Institution, Swan Lake